CLINICAL TRIAL: NCT05577403
Title: Effect of Mulligan's Mobilization With Movement Added With Isometric Exercises on Muscle Strength Pain and Disability Associated With Knee Osteoarthritis: A Randomized Controlled Study
Brief Title: Effect of Mulligans Mobilization With Movement in Osteoarthritis Knee.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Collaborators: King Saud University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RRC-2021-17
Record Dates: First submitted 2021-12-07; First posted 2022-10-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Knee
Keywords: Isometric exercise; Osteoarthritis; Rehabilitation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Mulligan's mobilization with movement added isometric strength training will be given 3 days a week for six weeks.
  Interventions: Behavioral: Mulligan's mobilization with movement MWM added isometric strength training
- Control Group (Active Comparator): Mobilization-added isometric strength training will be given 3 days a week for six weeks.
  Interventions: Behavioral: Mulligan's mobilization with movement MWM added isometric strength training

INTERVENTIONS:
Behavioral: Mulligan's mobilization with movement MWM added isometric strength training — Mulligan's mobilization with movement added isometric exercise:
  the participants in the experimental group will receive a Mulligan's mobilization with movement added isometric exercise.
  Treatment will be given for the period of three weeks, for five days a week in both groups.
  Data will be collected before intervention and after 2nd & 4th week of intervention.
  Other Names: Sham MWM added isometric strength training

SUMMARY:
To evaluate the effect of Mulligan's mobilization with movement in osteoarthritis of the knee.

DETAILED DESCRIPTION:
Patients with knee OA diagnosed at the orthopaedic clinic of Tumair general hospital and referred to the physiotherapy department who attended the rehabilitation centre of Majmaah university will be recruited.

Patients will be excluded if they have had a knee or hip injury, sensory deficits in the lower extremity, a history of lower-extremity surgery, a history of a quadriceps or hamstring muscle injury, low back-related leg pain, or any contraindication to manual therapy.

The protocol was submitted to and approved by the Rehabilitation Research Chair, King Saud University Research Ethics Committee (RRC-2021-17)

Participants will be requested to sign a written informed consent form approved by the institutional ethics committee. A total of 60 participants were randomly assigned to group A (experimental group): Mulligan's mobilization with movement MWM added isometric strength training, and group B (control group): Sham MWM added isometric strength training. Pre and post-test readings were taken at baseline, week 2, and week 4, respectively. The outcome measures for this study will be maximal voluntary isometric contraction of quadriceps strength (measured by ISOMOVE dynamometer), ROM, and Western Ontario and McMaster universities osteoarthritis (WOMAC) index.

ELIGIBILITY:
Inclusion Criteria:

* Patient with knee OA with radiological evidence of grade 2 or 3 of the Kellgren and Lawrence scale.
* Age between 40-65 years, unilateral or bilateral involvement (in the case of bilateral involvement, the more symptomatic knee was included), and pain in and around the knee.

Exclusion Criteria:

* Patient will be excluded, if they had any deformity of the knee, hip, or back, had any central or peripheral nervous system involvement.
* They had received steroids or intra-articular injection within the previous three months, uncooperative patients.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
pain intensity | 6 weeks
  Visual Analogue scale on 0 to10 cm
Range of Motion | 6 weeks
  Standard goniometer.
Western Ontario and McMaster universities osteoarthritis (WOMAC) index | 6 weeks
  Western Ontario and McMaster universities osteoarthritis scale

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan, PhD, Principal Investigator — Majmah University
Locations (1):
- Rehabilitation center, Majmaah University, Al Majma'ah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with the principal investigator (Dr. Shahnaz Hasan) and sub-investigator (Dr. Naiyer Shahzad) due to confidentiality issues.